CLINICAL TRIAL: NCT02906514
Title: Priming of Cardiopulmonary Bypass With Hydroxyethyl Starch 130/0.4 or Sodium Chloride 0.9% : a Double Blind Randomized Pilot Study in Adult Elective Conventional Cardiac Surgery
Brief Title: Priming of Cardiopulmonary Bypass With Hydroxyethyl Starch 130/0.4 or Sodium Chloride 0.9% : Pilot Study in Adult Elective Conventional Cardiac Surgery
Acronym: OPTIMUS-PRIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL15_0235
Record Dates: First submitted 2016-08-29; First posted 2016-09-20 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2018-02

CONDITIONS: Extracorporeal Circulation; Cardiac Surgery
Keywords: Hydroxyethyl Starch; Cardiac surgery; Priming of cardiopulmonary bypass
MeSH Terms: interventions — HES 130-0.4; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyethyl starch 130/0.4 (Experimental)
  Interventions: Drug: Non balanced Hydroxyethyl starch 130/0.4 (Voluven®, Fresenius)
- Sodium Chloride 0.9% (Placebo Comparator)
  Interventions: Drug: Sodium Chloride 0.9% (Fresenius)

INTERVENTIONS:
Drug: Non balanced Hydroxyethyl starch 130/0.4 (Voluven®, Fresenius) — 1000mL used for cardiopulmonary bypass priming
  Arms: Hydroxyethyl starch 130/0.4
Drug: Sodium Chloride 0.9% (Fresenius) — 1000mL used for cardiopulmonary bypass priming
  Arms: Sodium Chloride 0.9%

SUMMARY:
Best priming for cardiopulmonary bypass in cardiac surgery is unknown. Efficacy and toxicity of Hydroxyethyl Starch 130/0.4 used in this context are uncertain.

The aim of this pilot study is to determine if Hydroxyethyl Starch 130/0.4 is more effective than Sodium Chloride 0.9% in short term hemodynamic purpose without side renal or hemostatic effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective conventional cardiac surgery with cardiopulmonary bypass
* Patients insured under the French social security system

Exclusion Criteria:

* Pregnancy
* Patients placed under guardianship
* Urgent surgery
* Cardiac surgery without cardiopulmonary bypass
* Anterior cardiac surgery
* Non conventional cardiac surgery (mini-invasive surgery, dual valve replacement, right heart surgery)
* Simultaneous inclusion in another study with potential interference in outcomes
* Heparin-induced thrombocytopenia
* Chronic renal insufficiency (glomerular filtration rate < 60mL.min-1.m-2)
* Nature/nurture hemostasis disorders, in particular Von Willebrand disease and hemophilia
* Hydroxyethyl Starch allergy
* Weight under 33 kg
* Mechanical hemodynamic support at the end of the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Supplementary volume of fluid administered during cardiopulmonary bypass (ml) | Day 1 (From initiation to separation of cardiopulmonary bypass)
  Fluid administered during cardiopulmonary bypass for normal functioning, with the exception of blood product, cardioplegia and priming

SECONDARY OUTCOMES:
Variation of preoperative hematocrit and lowest hematocrit during cardiopulmonary bypass | Day 1 (From initiation to separation of cardiopulmonary bypass)
  Continuous monitoring of hematocrit during cardiopulmonary bypass.
Fluid balance | Hour 0
  Difference between total intraoperative volume of fluids administered (vascular filling, blood products, cardioplegia, priming) and total intraoperative volume of fluids loss (urine, bleedings)
Fluid balance | Hour 12
  Difference between total intraoperative volume of fluids administered (vascular filling, blood products, cardioplegia, priming) and total intraoperative volume of fluids loss (urine, bleedings)
Sequential Organ Failure Assessment score | Hour 24
Sequential Organ Failure Assessment score | Hour 0
Acid-Base parameters : arterial pH | Hour 24
Acid-Base parameters : Base Excess | Hour 0
Acid-Base parameters : Base Excess | H24
Acid-Base parameters : Lactatemia | Hour 0
Acid-Base parameters : Lactatemia | Hour 24
Acid-Base parameters : Chloremia | Hour 0
Acid-Base parameters : Chloremia | Hour 24
Coagulation parameters : platelets | Hour 0
Coagulation parameters : prothrombin | Hour 0
Coagulation parameters : activated partial thromboplastin | Hour 0
Coagulation parameters : fibrinogen level | Hour 0
Coagulation parameters : platelets | H24
Coagulation parameters : prothrombin | H24
Coagulation parameters : activated partial thromboplastin | H24
Coagulation parameters : fibrinogen level | H24
Hemoglobin level | Hour 0
Hemoglobin level | Hour 24
Surgical bleeding | Hour 12
Surgical bleeding | during surgical drainage, an average of 24 hours
Revision surgery for bleeding | Hour 12
Delay for ablation of surgical drainage | Day of ablation of surgical drainage, 24 hours
Antiemetic medication use | end of intensive care unit stay, 24 hours
  Any antiemetic medication used during this period
Delay to first extubation (number of hours) | Hour of first extubation, an average of 5 hours
Intensive care unit stay (number oh days) | Day of intensive care unit stay exit
Hospital stay (number of days) | Day of hospital exit, an average of 7 days
Creatinine level variation | Day 5
Creatinine level variation | Day 28
Creatinine level variation | Day 90
Renal replacement therapy use during intensive care stay | end of intensive care unit stay, an average of 24 hours
Renal replacement therapy dependency | Day 28
Renal replacement therapy dependency | Day 90
Mortality of any cause | During hospital stay, an average of 7 days
Mortality of any cause | Day 28
Mortality of any cause | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital Louis Pradel, Bron, France

REFERENCES:
- [Result] Schweizer R, Lameche M, Coelembier C, Portran P, Fornier W, Colombet B, Grinberg D, Pozzi M, Jacquet-Lagreze M, Fellahi JL. Cardiopulmonary Bypass Priming with Hydroxyethyl Starch 6% 130/0.4 or Sodium Chloride 0.9%: A Preliminary Double-Blind Randomized Controlled Study in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Dec;33(12):3534-3535. doi: 10.1053/j.jvca.2019.05.003. Epub 2019 May 10. No abstract available. PMID 31138465